CLINICAL TRIAL: NCT01348243
Title: MULTICENTRE, RANDOMIZED, OPEN-LABEL, TWO-ARM PARALLEL GROUPS, ACTIVE CONTROLLED STUDY DESIGN TO DEMONSTRATE EFFICACY AND TOLERABILITY OF CLODRONATE 200 MG/4 ML SOLUTION FOR INTRAMUSCULAR USE WITH 1% LIDOCAINE EVERY OTHER WEEK VS CLODRONATE 100 MG/3,3ML SOLUTION FOR INTRAMUSCULAR USE WITH 1% LIDOCAINE ONCE-WEEK IN A 1-YEAR TREATMENT PERIOD OF WOMEN WITH POSTMENOPAUSAL OSTEOPOROSIS
Brief Title: Efficacy Of Clodronate 200 Mg/4 Ml I.M. Solution With 1% Lidocaine Every Other Week Vs Clodronate 100 Mg/3,3ml I.M. Solution With 1% Lidocaine Once-Week In A 1-Year Treatment Period Of Women With Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC/PR/9900/004/10; 2010-022060-13 (EudraCT Number)
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Clodronic Acid; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clodronate 200 mg (Experimental)
  Interventions: Drug: disodium clodronate 200 mg/4 ml with 1% lidocaine
- Clodronate 100 mg (Active Comparator)
  Interventions: Drug: Disodium clodronate 100 mg/3,3 ml with 1% lidocaine

INTERVENTIONS:
Drug: disodium clodronate 200 mg/4 ml with 1% lidocaine — CLODRONATE 200 MG/4 ML SOLUTION FOR INTRAMUSCULAR USE WITH 1% LIDOCAINE EVERY OTHER WEEK
  Arms: Clodronate 200 mg
Drug: Disodium clodronate 100 mg/3,3 ml with 1% lidocaine — CLODRONATE 100 MG/3,3 ML SOLUTION FOR INTRAMUSCULAR USE WITH 1% LIDOCAINE ONCE-WEEK
  Arms: Clodronate 100 mg

SUMMARY:
Clodronic acid 100 mg/3,3 ml is used to prevent and treat postmenopausal osteoporosis.

The intramuscular formulation, which is given at a dose of 100 mg every 7 o 14 days, is at least as effective as daily oral therapy and appears more effective than intermittent intravenous treatment. Intramuscular clodronic acid in particular has also been associated with improvements in back pain. The drug is well tolerated, with no deleterious effects on bone mineralization, and use of parenteral therapy eliminates the risk of gastrointestinal adverse effects that may be seen in patients receiving oral bisphosphonates therapy.

In order to simplify the therapeutic dosing regimen, reducing the number of administrations per month, and therefore increase adherence to bisphosphonates therapy of the patient, a new formulation of disodium clodronic acid containing 200 mg/4 mL for i.m. administration has been developed. Lidocaine in this new formulation, as local anaesthetic, is maintained at the same concentration as in the 100 mg clodronic acid formulation.

The pharmacokinetics and tolerability of the intramuscular formulation of clodronic acid 200 mg in comparison to the marketed formulation clodronic acid 100 mg was evaluated in healthy post-menopausal volunteers. Two formulations were similar in terms of amount and rate of clodronic acid urinary excretion and in terms of safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedures;
2. Postmenopausal (any menses in the last 5 years) female subjects > 50 years old with lumbar or femoral-neck T-score < -2,5 and > -4;
3. At least three intact vertebrae between L1 and L4;
4. Patients treated according to the non-pharmacological standard of care;
5. Patients with the possibility and willingness to take the i.m. injections.

Exclusion Criteria:

1. BMI < 19 kg/m2;
2. History of: use of intravenous bisphosphonates, more than 12 months of bisphosphonates continuative or strontium ranelate use ever, or any use of bisphosphonates (oral and injective) within the last year, rhPTH use (recombinant human PTH) in the last 2 years, calcitonin use within the past 3 months, raloxifene and tamoxifen in the last 6 months or for more than 12 months in the last 2 years, fluoride (> 1 mg/die) for at least a month within the past 5 years;
3. Use of estrogen (oral or patch) for more than 1 month in the last 6 months or more than 12 months in the last 2 years;
4. Serious diseases of the oral cavity and surgery and/or dental implant from less than a month or planned in the next 12 months;
5. Type 1 or uncontrolled type 2 diabetes mellitus (defined as hemoglobin A1C >10,0), or currently using insulin;
6. Family history of malignant hyperthermia;
7. Heart disease, particularly bradyarrhythmias and heart failure; Adams-Stokes syndrome, Wolff-Parkinson-White syndrome or severe degrees of sinoatrial, atrioventricular or intraventricular block, acute cardiac decompensation;
8. History of kidney failure or renal insufficiency (serum creatinine > 2,0 mg/dl);
9. History of stroke in the last 6 months or uncontrolled hypertension;
10. Any history of hypercalciuria;
11. History of hypercalcemia, sarcoidosis, hyperparathyroidism, hypothyroidism or hyperthyroidism;
12. History of any malignancy except epithelioma considered cured ;
13. Patients currently treated with systemic prednisone or equivalent per day or > 2000 mcg beclomethasone dipropionate or equivalent daily; ;
14. Patients currently treated with antiepileptic drugs, anticoagulants or anticonvulsants or treated in the last 6 months or for more than 12 months in the last 2 years;
15. Patients current treated with propanolol, cimetidine or digitalis drugs;
16. History of alcohol or drug abuse;
17. Allergy, sensitivity or intolerance to study drugs (included lidocaine or other amide-type local anaesthetics) or excipients;
18. Subjects unlikely to comply with the study protocol or unable to understand the nature and scope of the study but also the possible benefits or unwanted effects of the study treatments;
19. Subjects who received any investigational new drug, or participated in clinical study within the last 12 weeks;
20. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Lumbar Bone Mineral Density | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico GB Rossi, Verona, Italy

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2010-022060-13